CLINICAL TRIAL: NCT06411912
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of NIDO-361 in Patients With Spinal and Bulbar Muscular Atrophy (SBMA)
Brief Title: A Study of NIDO-361 in Patients With SBMA
Acronym: PIONEER KD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nido Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDO-361-002
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Spinal and Bulbar Muscular Atrophy; Kennedy's Disease
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive NIDO-361 or placebo at the recommended Phase 2 dose (RP2D) of 100 mg once daily. Patients will receive daily oral doses of NIDO-361 or placebo for 12 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NIDO-361 (Experimental): Participants receive 100 mg of NIDO-361 given orally once daily.
  Interventions: Drug: NIDO-361
- Placebo (Placebo Comparator): Participants receive matched dose placebo given orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NIDO-361 — Tablets containing 100mg of NIDO-361 for oral administration.
  Arms: NIDO-361
Drug: Placebo — Placebo oral tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of NIDO-361 in adult patients with Spinal and Bulbar Muscular Atrophy (SBMA).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male
* Documented SBMA diagnosis confirmed by DNA genetic testing
* Able to complete six-minute walk test (6MWT)

Exclusion Criteria:

* Clinically significant cardiovascular, endocrine, hepatic, renal, pulmonary, gastrointestinal, neurologic, immunologic, malignant, metabolic, psychiatric, or other condition that, in the opinion of the Investigator, precludes the participant's safe participation in the study or would interfere with the study assessments
* Inability to undergo MRI (mild sedation may be allowed)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in thigh and total lean muscle volume as assessed by whole-body MRI | Through study completion, an average of 1 year
Number of patients with adverse events or serious adverse events. Number of patients discontinuing study and number of deaths. Number of mild, moderate, and severe adverse events. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- Rigshospitalet, Klinik for Nerve- og Muskelsygdomme & Copenhagen Neuromuscular Center, Copenhagen, Denmark
- Italy (2):
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedale Università di Padova, Padua
- Kyungpook National University Chilgok Hospital, Daegu, South Korea
- University of College London Hospital (UCLH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No